CLINICAL TRIAL: NCT06688656
Title: A Phase II Single-Center Exploratory Study on the Efficacy and Safety of Neoadjuvant Chemotherapy Sequentially Combined with Sintilimab in Resectable EGFR-Mutant Stage II-IIIB Non-Squamous Non-Small Cell Lung Cancer Patients
Brief Title: Neoadjuvant Chemotherapy Sequentially Combined with Sintilimab in Resectable EGFR-Mutant NSCLC
Acronym: Peri-E
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Hua Zhong, Dr., Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IS24145
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Lung Cancer
Keywords: NSCLC; EGFR; Neoadjuvant; Chemotherapy; PD-1
MeSH Terms: conditions — Lung Neoplasms | interventions — Pemetrexed; Carboplatin; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arm 1 (Other): Resectable EGFR-Mutant Stage II-IIIB Non-Squamous Non-Small Cell Lung Cancer Patients. Eligible subjects who meet the inclusion criteria and have signed the informed consent will receive sintilimab in combination with chemotherapy, with a treatment cycle of 3 weeks. A tumor assessment will be conducted before the start of the third cycle of treatment, and surgery will be performed within 3-6 weeks after the last cycle of neoadjuvant therapy, with a tumor assessment conducted 7 days prior to surgery. After completing local treatment (surgery), researchers will offer optional adjuvant therapy to patients, including EGFR-TKI.
  Interventions: Drug: Pemetrexed 500 mg/m2; Drug: carboplatin; Drug: Sintilimab

INTERVENTIONS:
Drug: Pemetrexed 500 mg/m2 — 1. Pemetrexed: 500mg/m² on Day 1, Q3W, administered via intravenous infusion for a total of 3 cycles.
Drug: carboplatin — AUC=5 on Day 1, Q3W，administered via intravenous infusion for a total of 3 cycles.
Drug: Sintilimab — Sintilimab, 200mg, administered via intravenous infusion on the 3rd day of each cycle, Q3W, for a total of 3 cycles.

SUMMARY:
This study is a prospective, single-arm, single-center Phase II trial, aiming to investigate efficacy and safety of neoadjuvant chemotherapy sequentially combined with sintilimab in resectable EGFR-mutant stage II-IIIB non-squamous NSCLC patients

DETAILED DESCRIPTION:
Previous studies have confirmed the efficacy of neoadjuvant chemotherapy and immunotherapy in NSCLC patients without driver gene mutations, while their effectiveness in patients with driver gene mutations remains controversial. This study is a prospective, single-arm, single-center Phase II trial targeting eligible subjects with resectable EGFR-mutated stage II-IIIB non-squamous non-small cell lung cancer, aiming to evaluate the efficacy and safety of sintilimab combined with chemotherapy as neoadjuvant therapy.

Eligible subjects who meet the inclusion criteria and have signed the informed consent will receive sintilimab in combination with chemotherapy, with a treatment cycle of 3 weeks. A tumor assessment will be conducted before the start of the third cycle of treatment, and surgery will be performed within 3-6 weeks after the last cycle of neoadjuvant therapy, with a tumor assessment conducted 7 days prior to surgery. After completing local treatment (surgery), researchers will offer optional adjuvant therapy to patients, including EGFR-TKI. Concurrently, dynamic blood samples will be collected before neoadjuvant therapy and after each treatment cycle for exploratory analysis, with the evaluation of MPR and pCR based on circulating tumor DNA minimal residual disease (ctDNA-MRD).

ELIGIBILITY:
Inclusion Criteria:

1. Sign a written informed consent prior to any study-related procedures;
2. Be aged ≥18 years;
3. Have a histopathologically confirmed diagnosis of stage II-IIIB (N2) non-squamous NSCLC, as per the9th edition TNM staging system by the International Association for the Study of Lung Cancer and the American Joint Committee on Cancer, with suspected N2 disease confirmed via mediastinoscopy or EBUS;
4. Have histologically, cytologically, or hematologically confirmed presence of EGFR-sensitive mutations (Ex19del, L858R), with co-existing driver mutations allowed;
5. Have sufficient tissue samples for PD-L1 immunohistochemistry and NGS mutation testing; if tissue samples are inadequate, consent to undergo blood NGS testing;
6. PD-L1 expression level ≥1%;
7. Have at least one radiologically measurable lesion as per the RECIST criteria version1.1;
8. Be assessed by a surgeon as having pulmonary or other organ function sufficient to tolerate local surgical treatment;
9. Have no prior history of anti-tumor treatment;
10. Have an ECOG performance status of0-1;
11. Have an expected survival time >3 months;
12. Possess adequate organ function, meeting the following laboratory criteria: a) Absolute neutrophil count (ANC) ≥1.5x10^9/L without the use of granulocyte colony-stimulating factor within the past14 days; b) Platelets ≥100x10^9/L without transfusion within the past14 days; c) Hemoglobin >9g/dL without transfusion or use of erythropoiesis-stimulating agents within the past14 days; d) Total bilirubin ≤1.5 times the upper limit of normal (ULN); e) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 times ULN (ALT or AST ≤5 times ULN allowed in subjects with liver metastases); f) Creatinine ≤1.5 times ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥60 ml/min; g) Adequate coagulation function, defined as an international normalized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN; h) Normal thyroid function, defined as thyroid-stimulating hormone (TSH) within normal range. Subjects with baseline TSH outside the normal range may be included if total T3 (or FT3) and FT4 are within normal limits; i) Cardiac enzymes within normal range (isolated laboratory abnormalities deemed clinically insignificant by the investigator may also be included);
13. For female subjects of childbearing potential, a negative urine or serum pregnancy test must be obtained within3 days prior to the first administration of the study drug (Day1 of Cycle1). If the urine pregnancy test is inconclusive, a blood pregnancy test is required. Non-childbearing potential is defined as being post-menopausal for at least one year, surgically sterilized, or having undergone a hysterectomy;
14. All subjects (both male and female) at risk of conception must agree to use a highly effective method of contraception with a failure rate of less than1% throughout the treatment period and for120 days (or180 days) after the last administration of the study drug.

Exclusion Criteria:

1. Pathology of small cell lung cancer (SCLC), including mixed SCLC and NSCLC;
2. Stage I and IV NSCLC, patients who have previously received systemic antitumor treatments such as immunotherapy, targeted therapy, or chemotherapy;
3. Stage III unresectable NSCLC patients;
4. Patients with rare EGFR mutations;
5. Diagnosis of any malignancy other than NSCLC within5 years prior to the first dose, excluding adequately treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or carcinoma in situ that has been surgically cured;
6. Currently participating in an interventional clinical study or having received other investigational drugs or device therapies within4 weeks prior to the first dose;
7. Use of traditional Chinese medicine or immunomodulatory drugs with indications for NSCLC within2 weeks prior to the first dose (including thymosin, interferon, interleukin, except for local use to control pleural effusion);
8. Active autoimmune disease requiring systemic treatment (such as disease-modifying drugs, corticosteroids, or immunosuppressants) within2 years prior to the first dose; replacement therapy (e.g., thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) is not considered systemic treatment;
9. Systemic corticosteroid therapy (excluding nasal, inhaled, or other local routes of corticosteroid administration) or any other form of immunosuppressive therapy within7 days prior to the first dose; Note: Physiological doses of corticosteroids (≤10 mg/day of prednisone or equivalent) are permitted;
10. Clinically uncontrollable pleural effusion/ascites (subjects who do not require drainage or whose effusion does not significantly increase after stopping drainage for3 days may be enrolled);
11. Known history of allogeneic organ transplantation (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
12. Known allergy to study drugs such as sintilimab, pemetrexed, carboplatin, their active ingredients, or excipients;
13. Inadequate recovery from toxicity and/or complications from any prior intervention before starting treatment (i.e., ≤ Grade1 or back to baseline, excluding fatigue or alopecia);
14. Known history of human immunodeficiency virus (HIV) infection (i.e., positive for HIV1/2 antibodies);
15. Untreated active hepatitis B (defined as positive for HBsAg and detected HBV-DNA copy number exceeding the upper limit of normal of the testing laboratory at the study center); Note: Hepatitis B subjects meeting the following criteria may also be enrolled: a) HBV viral load <1000 copies/ml (200 IU/ml) before the first dose, and the subject should receive anti-HBV treatment throughout the chemotherapy period to prevent viral reactivation; b) For subjects who are anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-), prophylactic anti-HBV treatment is not required, but close monitoring for viral reactivation is necessary;
16. Active HCV infection (positive for HCV antibodies and HCV-RNA levels above the detection limit);
17. Vaccination with a live vaccine within30 days prior to the first dose (Day1, Cycle1); Note: Administration of an injectable inactivated virus vaccine for seasonal influenza is allowed within30 days prior to the first dose, but administration of a live attenuated influenza vaccine via nasal route is not permitted;
18. Pregnant or breastfeeding women;
19. Presence of any severe or uncontrolled systemic disease, such as: a) Significant and symptomatically severe abnormalities in rhythm, conduction, or morphology on resting electrocardiogram, such as complete left bundle branch block, second-degree or higher heart block, ventricular arrhythmias, or atrial fibrillation; b) Unstable angina, congestive heart failure, chronic heart failure of NYHA class ≥2; c) Myocardial infarction within6 months prior to enrollment; d) Uncontrolled blood pressure (systolic >140 mmHg, diastolic >90 mmHg); e) History of non-infectious pneumonia requiring corticosteroid treatment within1 year prior to the first dose, or current clinically active interstitial lung disease; f) Active pulmonary tuberculosis; g) Active or uncontrolled infection requiring systemic treatment; h) Clinically active diverticulitis, intra-abdominal abscess, gastrointestinal obstruction; i) Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis; j) Poorly controlled diabetes (fasting blood glucose (FBG) >10mmol/L); k) Urinalysis indicating proteinuria ≥++, and confirmed24-hour urinary protein quantification >1.0 g; l) Presence of psychiatric disorders that may interfere with treatment compliance;
20. Any history, disease evidence, treatment, or laboratory test abnormalities that might interfere with the results of the trial, hinder full participation in the study, or other conditions deemed inappropriate for enrollment by the investigator, or potential risks considered by the investigator as unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-31 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
major pathological response (MPR) | Evaluated within 2 weeks post-surgery.
  MPR is defined as ≤10% residual viable tumor cells in the lung and lymph nodes, to be evaluated within 2 weeks post-surgery.

SECONDARY OUTCOMES:
Pathological Complete Response (pCR) | Evaluated within 2 weeks post-surgery.
  pCR is defined as the absence of residual tumor in both the lung and lymph nodes after neoadjuvant therapy
Event-Free Survival (EFS) | up to 3 years after enrollment
  EFS is defined as the time from the start of neoadjuvant therapy to the occurrence of any disease progression that precludes surgery, post-surgical disease progression or recurrence, disease progression without surgery, or death from any cause. It is measured from the start of neoadjuvant therapy to the first recorded date of disease progression or death (whichever occurs first).

CONTACTS AND LOCATIONS:
Locations (1):
- 241, West Huaihai Road, Shanghai, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No